CLINICAL TRIAL: NCT06447545
Title: Comparison Between Low Pressure Pneumoperitoneum with High Pressure Pneumoperitoneum in Post-operative Pain, Shoulder Tip Pain and Common Bile Duct Injuries in Patients Undergoing Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulab Devi Hospital (Other)
Responsible Party: Principal Investigator, Zain Himayoun, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAMC/IRB/EA 31 2024
Record Dates: First submitted 2024-05-24; First posted 2024-06-07 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-06

CONDITIONS: Cholecystectomy; Pneumoperitoneum; Pain, Postoperative
MeSH Terms: conditions — Pneumoperitoneum; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Pressure Pneumoperitoneum (Other): low-pressure pneumoperitoneum in which the pressure is (6-10 mmHg)
  Interventions: Device: Changing pressure of Pneumoperitoneum to 6-10 mmHg
- High Pressure Pneumoperitoneum (Other): High-pressure pneumoperitoneum, involving insufflation pressures typically ranging from 12 to 15 mmHg or higher
  Interventions: Device: Changing pressure of Pneumoperitoneum to 12-15 mmHg

INTERVENTIONS:
Device: Changing pressure of Pneumoperitoneum to 6-10 mmHg — Result of changing pneumoperitoneum pressure on CBD injury and pain
  Other Names: Low Pressure Pneumoperitoneum
  Arms: Low Pressure Pneumoperitoneum
Device: Changing pressure of Pneumoperitoneum to 12-15 mmHg — Result of changing pneumoperitoneum pressure on CBD injury and pain
  Other Names: High Pressure Pneumoperitoneum
  Arms: High Pressure Pneumoperitoneum

SUMMARY:
This study aims to address the existing gap in knowledge by conducting a comprehensive comparison of the incidence of pain and common bile duct injuries in patients undergoing laparoscopic cholecystectomy using Low pressure pneumoperitoneum versus high pressure pneumoperitoneum.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is minimally invasive surgery to remove the gallbladder. It helps people when gallstones cause inflammation, pain or infection. Since the early 1990s, the laparoscopic cholecystectomy technique has largely supplanted the open approach for routine gallbladder removal. This method is recommended for various conditions such as cholecystitis (both acute and chronic), symptomatic cholelithiasis, biliary dyskinesia, acalculous cholecystitis, gallstone pancreatitis, and gallbladder masses/polyps-similar to the indications for an open cholecystectomy. Gallbladder cancers, however, are typically better addressed through open cholecystectomy. In the United States, around 20 million people have gallstones, leading to approximately 300,000 cholecystectomies annually. Ten to fifteen percent of the population has asymptomatic gallstones, and among them, 20% experience symptoms such as biliary colic. Complications, including acute cholecystitis, gallstone pancreatitis, choledocholithiasis, and gallstone ileus, manifest in approximately 1% to 4% of symptomatic cases. Gallstone prevalence increases with age, with women between 50 to 65 years having a 20% incidence, compared to 5% in men. Cholesterol constitutes 75% of gallstones, while the remaining 25% are pigmented; however, clinical signs and symptoms remain consistent regardless of the gallstone composition.1 Low-pressure and high-pressure pneumoperitoneum, both integral to laparoscopic cholecystectomy, have been subjects of extensive research, primarily focusing on their impact on post-operative pain management.

Traditionally, in laparoscopic cholecystectomy, one of the initial procedures involves creating pneumoperitoneum. This is done by introducing carbon dioxide (CO2) either through a veress needle or a port in the abdominal wall. The CO2 is then gently infused into the peritoneal cavity, reaching a pressure of 10-20 mmHg, at a rate of 4-6 litres per minute. To maintain the pneumoperitoneum, a steady gas flow of 200-400 ml/min is sustained. In conventional laparoscopic cholecystectomy, a higher intra-abdominal pressure of 12-15mmHg is used, while low-pressure pneumoperitoneum laparoscopic cholecystectomy employs pressures below 8mmHg.2 High-pressure pneumoperitoneum, involving insufflation pressures typically ranging from 12 to 15 mmHg or higher, facilitates enhanced intraoperative visualization, ease of surgical manipulation, and shorter operative times. However, despite these advantages, it commonly correlates with increased post-operative pain and discomfort, particularly in the form of referred shoulder pain. The mechanism behind this pain is attributed to diaphragmatic irritation and irritation of the phrenic nerve due to the increased pressure within the peritoneal cavity.3 In contrast, low-pressure pneumoperitoneum, characterized by lower insufflation pressures, often ranging from 8 to 12 mmHg, aims to mitigate the post-operative discomfort experienced by patients. Studies exploring the use of lower pressures have indicated promising outcomes in reducing post-operative pain levels, shoulder discomfort, and overall patient discomfort following laparoscopic cholecystectomy.4 Although low-pressure pneumoperitoneum may potentially prolong the operative duration due to decreased visibility and the need for more delicate surgical manoeuvres, it presents a viable option for patients prone to experiencing heightened post-operative pain. The advantages of decreased pain, reduced shoulder discomfort, and potentially faster recovery post-surgery make low-pressure pneumoperitoneum an appealing consideration, especially for patients with a lower threshold for pain or those with a history of difficulties in managing post-operative discomfort. According to recent study pain was experienced in 22.5 % in Low pressure vs 57% in high pressure pneumoperitoneum technique 5,6

Bile duct injury (BDI) following cholecystectomy, particularly laparoscopic cholecystectomy (LC), is indeed a serious complication associated with significant morbidity and mortality. The incidence of BDI has increased with the adoption of laparoscopic techniques. The complications often result from anatomical misperceptions or inadvertent dissection, leading to injury to the common bile duct (CBD). Several factors contribute to the increased incidence of BDI in LC compared to open cholecystectomy. These include disorientation of anatomical variables, inadvertent dissection at Calot's triangle, or visual misperception by the operating surgeon. Proximal injuries, occurring within 2cm from the bifurcation, are becoming more prevalent. Recognition of CBD injury is crucial for prompt and effective management, as delayed diagnosis can lead to severe complications such as systemic inflammatory response syndrome and multi-organ failure syndrome. The time of presentation of these injuries can vary, making early detection challenging. Preventing common bile duct injury involves several key principles:

1. Optimal Exposure of Calot's Triangle: Proper exposure of Calot's triangle allows the surgeon to visualize the anatomical structures clearly, reducing the risk of inadvertent injury.
2. Judicious Use of Diathermy Near CBD Territory: Careful use of diathermy (electrosurgery) near the CBD is essential to avoid thermal injury. Excessive use of diathermy can lead to tissue damage and increase the risk of bile duct injury.
3. Use of a 30-Degree Telescope: A 30-degree laparoscope provides a better angle of vision, enhancing the surgeon's ability to visualize anatomical structures accurately during laparoscopic procedures.
4. Safe Clip Application without Tenting of CBD: Applying clips to secure structures without tenting the CBD helps avoid compression and potential injury. Proper clip placement is crucial for securing structures while minimizing the risk of damage to nearby tissues.
5. Adherence to the Rule of Thumb: Surgeons should be mindful of the "rule of thumb" to prevent common bile duct injury. This involves meticulous and precise surgical technique, including gentle tissue handling and avoiding excessive traction on the structures.

In conclusion, preventing common bile duct injury during cholecystectomy requires a combination of technical skill, anatomical knowledge, and adherence to established principles. Surgeons must be vigilant and adopt a cautious approach to minimize the risk of this serious complication. Early recognition and active management of CBD injuries are essential for improving patient outcomes and reducing morbidity and mortality associated with this iatrogenic catastrophe7.

The choice between these techniques involves a careful consideration of multiple factors, including the specific characteristics of the patient, the surgeon's expertise, and the complexities of the surgical procedure. As medical practitioners continue to explore ways to enhance patient outcomes and minimize post-operative discomfort, the debate between low-pressure and high-pressure pneumoperitoneum in laparoscopic cholecystectomy remains an active area of research and clinical consideration.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both genders
* Patients undergoing laparoscopic cholecystectomy for cholelithiasis.

Exclusion Criteria:

* Patients with cardiac abnormalities.
* Patients with previous abdominal surgeries.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of pain and common bile duct injury in patients undergoing laparoscopic cholecystectomy using Low pressure pneumoperitoneum is less versus High pressure pneumoperitoneum. | 6 months
  Pain will accessed using VAS. Pain (VAS): The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). It was assessed at 4, 8, 12 hours post-operatively by using Visual Analogue Pain Scale.
  No pain |0____1____2____3____4____5____6____7____8____9____10| sever pain Mild pain-Moderate Pain-Sever pain Visual Analogue Pain Scale And CBD injury will be accessed using bismuth classification.
  CBD INJURY: Injury to CBD Is Classified According to Bismuth Classification:
  Type I is a low injury with a stump length more than 2 cm. Type II is a middle level injury with a stump length less than 2 cm. Type III is a high-level injury without common hepatic duct available but preserved confluence.
  Type IV involves loss of hepatic confluence with no communication between right and left ducts.

CONTACTS AND LOCATIONS:
Overall Officials: M. Zia-ul-Miraj Ahmad, MBBS,FRCS, Study Director — Gulab Devi Hospital
Locations (1):
- Gulab Devi Hospital, Lahore, PUN, Pakistan